CLINICAL TRIAL: NCT03253484
Title: Laser Treatment in Early Wound Healing to Promote Physiological Skin Remodeling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Katrine Elisabeth Karmisholt, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-17012492
Record Dates: First submitted 2017-08-11; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Scar Improvement by Laser
Keywords: scar NAFL laser

STUDY DESIGN:
Intervention Model Description: split scar study
Who Masked: Outcomes Assessor
Masking Description: the outcome assessor will not know which side is the treated side of scar
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAFL-treated wounds (Experimental): NAFL treated wounds
  Interventions: Radiation: NAFL-treatment
- Control (No Intervention): untreated control wound

INTERVENTIONS:
Radiation: NAFL-treatment — non ablative fractional laser 15 40 nm promoting wound healing and reduction of scar formation
  Arms: NAFL-treated wounds

SUMMARY:
The primary objective of this study is to explore the potential clinical effect of targeting surgical wounds in all three wound healing phases by non ablative fractional laser (NAFL) to reduce scar formation in a randomized controlled trial. Thus, NAFL will be applied during 1) inflammation phase (0-3 days) as represented by NAFL-treatment adjacent to surgical wounding, 2) proliferation phase (4-21 days) by NAFL-treatment immediately after suture removal and 3) remodeling phase (21 days-1 year) by NAFL-treatment six weeks after surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, assessor - blinded, intra-individual trial comparing laser exposed skin lesions to untreated control skin lesions in a split scar set-up to investigate efficacy. The study will be performed on patients undergoing an excision at Bispebjerg Dermatological Department. One randomly allocated part of each included wound will receive three NAFL-treatments and the other part will serve as untreated control wound. Scars will be evaluated clinically on-site by blinded evaluator immediately before third treatment and 3 months after NAFL-treatments. The clinical data will be supplemented by blinded photo-evaluation, patients' evaluation and non-invasive measurements.

ELIGIBILITY:
Inclusion Criteria:

* o Subjects referred to excision of either benign, pre malignant or malignant non-melanoma skin cancer (NMSC) lesions.

  * The length of postoperative wound should be estimated to minimum 2.5 cm and may be located on any region of the body
  * Minimum 18 years old
  * Presenting full medical record report at study initiation
  * Fitzpatrick skin type I-III
  * Non-smokers
  * Written informed consent obtained from subject
  * Understanding of investigation procedures and willingness to abide to all procedures during the course of the investigation

Exclusion Criteria:

* o History of or presenting with a keloid scar

  * A subject with a systemic disease not yet stabilized
  * If the patient is pregnant
  * Visible recent sun exposure in test area
  * Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study
  * Current use of topical treatment and lack of willingness to refrain from future use of topical treatment, such as i.e. silicone products, that potentially can interfere with the test results
  * Unable to follow the outlined study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-08-18 (Estimated); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Clincial evaluation on Patient observer scar assessement scale (POSAS) | 3 months followup
  validated scar scale

SECONDARY OUTCOMES:
Photoevaluation on visual analogue scale | 3 months follow-up
  3 independent dermatologists will evaluate on VAS
Reflectance measurement | 3 months followup
  measurement of erythema and pigment
Clinical evaluation on Vancouver Scar Scale | 3 months followup
  validated scar scale
Clincial evaluation on Patient observer scar assessement scale (POSAS) | 1month follow-up
  validated scar scale
Clinical evaluation on Vancouver Scar Scale | 1month follow-up and
  validated scar scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karmisholt KE, Banzhaf CA, Glud M, Yeung K, Paasch U, Nast A, Haedersdal M. Laser treatments in early wound healing improve scar appearance: a randomized split-wound trial with nonablative fractional laser exposures vs. untreated controls. Br J Dermatol. 2018 Dec;179(6):1307-1314. doi: 10.1111/bjd.17076. Epub 2018 Sep 30. PMID 30101519